CLINICAL TRIAL: NCT06438276
Title: Supporting Adolescent Mental Health by Psychiatric Outreach Nurses: A Mixed Method Evaluation Study
Brief Title: Psychiatric Outreach Nurses Supporting Adolescent Mental Health
Acronym: JAPSY
Status: Recruiting | Type: Observational
Sponsor: University of Eastern Finland (Other)
Collaborators: Wellbeing Services County of North Savo (Unknown); The Foundation for Municipal Development (Unknown)
Responsible Party: Sponsor
Other Study IDs: JAPSY_20230
Record Dates: First submitted 2024-05-06; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Depression; Anxiety
Keywords: mental health; mental disorders; adolescent; outreach service; school-based; effectiveness; economic evaluation
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being; Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolescents with mood disorders seeking help in student welfare services: Intervention group receiving psychiatric outreach nurse services: adolescents (12-16 years old) who seek help from student welfare services due to mood disorders and have access to psychiatric outreach nurse's service.
  Control group receiving TAU: adolescents (12-16 years old) who seek help from student welfare services due to mood disorders and have no access to psychiatric outreach nurse's service.
  Interventions: Behavioral: Psychiatric outreach nurse service

INTERVENTIONS:
Behavioral: Psychiatric outreach nurse service — Mental health service provided by psychiatric outreach nurses for 12-16 year old students in secondary schools

SUMMARY:
The study evaluates the effectiveness and cost-effectiveness of the outreach work of psychiatric registered nurses (RN) and the experiences of professionals in the field. The service is provided in school environment. First, the study will assess the effectiveness of brief interventions provided by psychiatric outreach nurses on the perceived mental health and quality of life of adolescents (12-16 year old pupils) and their use of social and health services, compared to the support/treatment provided by conventional student welfare services at 6 and 12 months follow-up. The intervention is an outreach service provided by psychiatric nurses. In the intervention, the psychiatric registered nurse will implement interventions such as usual care, discussion, psychoeducation, substance abuse skills and various methods (such as interpersonal psychotherapy = IPT-N and Cool Kids) and motivational interviewing.

Secondly, an economic evaluation of the service will be carried out at 6 and 12 months follow-up. The economic evaluation will be carried out from the perspective of the Wellbeing Services County, including the costs of implementing the intervention model and its effects on adolescents' use of student welfare services as well as other social and health services. Primarily, the economic evaluation will use quality-weighted life years as a measure of effectiveness. Also analysis using depression, anxiety and substance use measures will be conducted. Thirdly, the study will explore the experiences of psychiatric nurses implementing the service as well as the experiences of their collaborators in schools (public health nurses, school social workers, psychologists, doctors and teachers) about the service and its implementation.

DETAILED DESCRIPTION:
Quantitative research data will be used to evaluate the effectiveness of the psychiatric outreach care compared to conventional care (TAU). Psychiatric outreach registered nurses are currently available in some schools in several municipalities in the North Savo region in Finland. In the other schools, support is provided by so-called "usual" counselling and other support/treatment, e.g. by public health nurses, school social workers, school psychologists and school doctors.

The study design is a clustered controlled setting. The target sample size for quantitative data is 160 participants. The intervention group (n = 80) will consist of pupils receiving support/treatment from psychiatric outreach nurses. The control group (n = 80) will consist of pupils whose schools provide standard student welfare services and whose mental health status and support needs are similar to those of the intervention group.

The data will be collected through questionnaires administered to secondary school pupils to assess their mental health status and quality of life. The adolescents' service use in terms of student welfare services as well as Wellbeing Services County's social and health care services will be collected through questionnaires. At baseline, the use of services will be surveyed retrospectively over a six-month period.

The primary outcome variable of the intervention is the adolescent's perceived mental health status as assessed by the PHQ-9-A (Patient Health Questionnaire) measure of depression and the GAD-7 (generalized anxiety disorder) measure of anxiety. The secondary outcome variables are the adolescent's perceived quality of life (EQ-5D-Y, five dimensional quality of life measure) and substance use (ADSUME, Adolescents´ Substance Use Measurement). The study will primarily investigate the effect of psychiatric outreach nurses on treatment response. Secondarily, subgroups of at least 20 participants will be examined (e.g. controls for gender, age or other background variables).

Participants are assigned to the intervention or control group based on whether the services of an psychiatric outreach nurse is available in their school (intervention) or not (control).

For similarities and differences between the intervention and control groups, a descriptive analysis is performed using the chi-square test to compare categorical variables and the t-test or Mann-Whitney U-test to compare continuous variables. The effectiveness of the intervention will be analysed using statistical methods appropriate for panel data, taking into account the effects of possible correlation/multicollinearity on the results. Statistical methods will be used to control for the possible selection of a non-standardised design by including control variables in the models.

The economic evaluation of the intervention will use data on the use of social and health services, student welfare services and the cost of the intervention. Data on the costs of the intervention will be obtained from the Wellbeing Services County of North Savo. The costs of health and social services and student welfare services are calculated on the basis of the number of services used and the unit costs. The cost-effectiveness of the intervention is analysed in relation to the treatment as usual provided by student welfare services using incremental net monetary benefit or incremental net health benefit evaluation to examine differences in costs and/or health benefits between groups and in the above-mentioned outcomes at 6-month and 12-month follow-up. Primarily, the economic evaluation will use the EQ-5D-Y measure to calculate quality-weighted life-years. In addition, the results of the PHQ-9-A, GAD-7 and ADSUME measures will be analysed.

Eligibility Criteria: Pupils (12-16 years old) who seek help from a student welfare service due to mood disorders. In addition, a representative of the student welfare service (e.g. a public health nurse, school social worker, psychologist or doctor) or a representative of the student welfare service and an psychiatric outreach nurse assess together a person's eligibility for the study, taking into account the inclusion and exclusion criteria.

Inclusion criteria for the intervention and control groups will be one or more of the following symptoms: prolonged and/or complicated anxiety, mood symptoms, obsessive-compulsive and/or eating disorder symptoms, mild to moderate self-harm (e.g. death wishes or cutting). In addition, the young person's motivation to receive the service is an admission criterion.

Exclusion criteria: The psychiatric outreach nurse service is not suitable for persons with one or more of the following needs or life situations: pupils who need light support and guidance, young people with a single problem of low motivation for school, young people with a stressful life situation or relationship problems. On the other hand, the service is not intended for pupils who are in acute need of specialist care or for pupils with multidisciplinary problems for whom support measures have already been put in place, because of their mental health symptoms (e.g. severe depression, psychotic symptoms, severe and acute suicidal tendencies or a clear suicide plan). Exclusion criteria for the intervention and control groups also include situations where the young person has a long-lasting, already established mental health problem and/or a need for further treatment after a period of specialised hospital care. Exclusion criteria also include behavioural disorders where there is a clear underlying cause other than a mental disorder.

The qualitative perspective of the study focuses on those implementing the service (psychiatric outreach nurses) and their collaborators in schools (e.g. school social workers, public health nurses, school psychologists, doctors and teachers). The total number of interviewees is estimated to be 15-20. Data collection consists of individual semi-structured interviews to describe the interviewees' experiences of applying the new service approach in the school setting. As the approach is new in the Wellbeing Services County of North Savo, it is necessary to explore the experiences of both those implementing as well as their collaborators in terms of introducing the service, operation of the service, the perceived needs for the service as well as the needs for development of the service. The interviews will be carried out at the beginning of the study and at 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents (12-16 years old) who seek help from student welfare services due to mood disorders and who have one or more of the following conditions: prolonged and/or complicated anxiety, mood symptoms, obsessive-compulsive and/or eating disorder symptoms, mild to moderate self-harm (e.g. death wishes or cutting). In addition, person's motivation to receive the service provided is an admission criterion.

Exclusion Criteria:

* Persons with one or more of the following needs or life situations: adolescents who need light support and guidance, young people with a single problem of low motivation for school, young people with a stressful life situation or relationship problems. On the other hand, adolescents who are in acute need of specialist care or for adolescents with multidisciplinary problems for whom support measures have already been put in place, because of their mental health symptoms (e.g. severe depression, psychotic symptoms, severe and acute suicidal tendencies or a clear suicide plan).
* Exclusion criteria for the intervention and control groups also include situations where the adolescent has a long-lasting, already established mental health problem and/or a need for further treatment after a period of specialised hospital care.
* Exclusion criteria also include behavioural disorders where there is a clear underlying cause other than a mental disorder.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Adolescent (12-16 year old) students of secondary schools in the municipalities of North Savo Wellbeing County who seek help from student welfare services due to mood disorders.
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire modified for adolescent to measure perceived mental health | 6-month and 12-month follow-up
  The effects of the outreach psychiatric nurse service on adolescent's perceived mental health status assessed by the Patient Health Questionnaire modified for adolescent (PHQ-9-A) measure of depression in 6-month and 12-month follow-up. The minimum value of the measure is 0 and maximum value 27. Higher scores is worse outcome.
Generalized Anxiety Disorder 7-item to measure adolescent's perceived mental health | 6-month and 12-month follow-up
  The effects of the outreach psychiatric nurse service on adolescent's perceived mental health status assessed by the Generalized Anxiety Disorder 7-item (GAD-7) measure of anxiety in 6-month and 12-month follow-up. The minimum value of the measure is 0 and maximum value 21. Higher scores is worse outcome.

SECONDARY OUTCOMES:
EuroQol-5-Dimension 3-Level modified for adolescent to measure perceived quality of life | 6-month and 12-month follow-up
  The effects of the outreach psychiatric nurse service on adolescent's perceived quality of life and substance use assessed by EuroQol- 5-Dimension 3-Level modified for adolescent (EQ-5D-Y-3L) measure in 6-month and 12-month follow-up. EQ-5D-Y will be converted to index-values [theoretical range 0-1] by using suitable value set. The higher value means better health related quality of life.
Adolescents' Substance Use Measurement to measure substance use | 6-month and 12-month follow-up
  The effects of the outreach psychiatric nurse service on adolescent's substance use assessed by Adolescents' Substance Use Measurement (ADSUME) measure in 6-month and 12-month follow-up.The minimum value of the measure is 0 and maximum value 90. Higher scores is worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Lammintakanen, PhD, Professor, Principal Investigator — University of Eastern Finland
Locations (1):
- Wellbeing Services County of North Savo, Kuopio, Northern Savonia, Finland

IPD SHARING:
Plan to Share IPD: No